CLINICAL TRIAL: NCT03495180
Title: Quantitative SSEP and EEG As Objective Pain Biomarker
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Froelich, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 67890123
Record Dates: First submitted 2018-03-27; First posted 2018-04-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard EEG or SSEP (Experimental): the intensity of an experimental pain stimulus and perceived (self-rating, subjective) pain intensity.
  Interventions: Other: Standard EEG or SSEP

INTERVENTIONS:
Other: Standard EEG or SSEP — The gamma frequency range (30 -100 Hz) of standard EEG or somatosensory evoked potential (SSEP) correlate with intensity of an experimental pain stimulus and perceived (self-rating, subjective) pain intensity.

SUMMARY:
Over the past few years, significant advances have begun to be made in the development of particular measures as valid biomarkers or surrogate markers for the presence of acute and chronic pain. Many of these advances have been made because of the development of new and improved technologies, for example in the fields of imaging and genetics. Research is now showing brain activity and brain organizational changes associated with the presence of pain. Various factors have been found in the blood that is associated with the presence of pain. Research is also suggesting that pupil responses to a variety of stimuli may predict the presence of pain. And machine learning analysis of videos has found facial movement patterns in both animals and humans that are correlated with the presence of pain.

This is a pilot study to investigate whether components of a person's electrical brain activity do reflect pain sensation.

DETAILED DESCRIPTION:
Over the past few years, significant advances have begun to be made in the development of particular measures as valid biomarkers or surrogate markers for the presence of acute and/or chronic pain. Many of these advances have been made because of the development of new and improved technologies, for example in the fields of imaging and genetics. Research is now showing brain activity and brain organizational changes associated with the presence of pain. Various factors have been found in the blood that is associated with the presence of pain. Research is also suggesting that pupil responses to a variety of stimuli may predict the presence of pain and machine learning analysis of videos has found facial movement patterns in both animals and humans that are correlated with the presence of pain.

The establishment of a biomarker of pain is a key requirement for understanding the person-specific effects of anesthetic and analgesic drugs. An objective pain measure will be an integral part in the planning of an anesthetic and potentially enable the researchers to answer the question whether proper matching of the anesthetic or analgesic dose to a person's individual profile will result in better cognitive recovery from anesthesia.

There are several approaches to quantifying pain in an objective fashion. These approaches are based on the observation of afferent signals to the brain, brain integration of nociceptive signals or secondary responses to nociceptive signals (ocular, facial, autonomic or behavioral responses). Pain has been studied extensively with fMRI. Several other methods have been proposed: pain behavior, pupillary responses, and autonomic responses.

Somatosensory evoked electrical potentials (SSEP) are routinely recorded to assess the integrity of sensory pathways during spine surgery. Our primary study aim is to correlate the neuronal (EEG) signal (Y1) and/or γ - band power (Y2) with both the stimulus intensity (X1, the voltage of constant current stimulator output) and the perceived pain intensity (X2)

This is a pilot study to test the hypothesis that the gamma frequency range (30 -100 Hz) of standard EEG or somatosensory evoked potential (SSEP) correlate with intensity of an experimental pain stimulus and perceived (self-rating, subjective) pain intensity.

.

ELIGIBILITY:
Inclusion Criteria:

* Adult human volunteers (age > 18) that are able to understand study procedures.

Exclusion Criteria:

* Medical conditions that would interfere with somatosensory processing. (diabetic neuropathy, stroke), chronic pain, medications known to affect pain processing (opioid therapy, selective serotonin reuptake inhibitor (SSRI)).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of (electrical) pain intensity (X) and amplitude of SSEP (Y). | 20 minutes during the study session (once).
  Pearson Correlation of X and Y.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Froelich, MD, Principal Investigator — UAB Department of Anesthesiology, Critical Care Division

IPD SHARING:
Plan to Share IPD: Undecided